CLINICAL TRIAL: NCT02670902
Title: Intervention for Persons With Co-Occurring Disorders Leaving Residential Tx
Brief Title: Intervention for Persons Leaving Residential Substance Abuse Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K01DA035330 (NIH)
Record Dates: First submitted 2016-01-25; First posted 2016-02-02 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-05

CONDITIONS: Substance Use Disorders
Keywords: Residential substance use treatment; Transition
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Critical Time Intervention-Residential (Experimental): CTI-R is a 9-month, assertive outreach and linkage program.
  Interventions: Behavioral: Critical Time Intervention-Residential (CTI-R); Behavioral: Enhanced Usual Discharge Services-Residential
- Enhanced Usual Discharge-Residential (Active Comparator): The enhanced usual discharge condition includes usual discharge services plus enhanced transition services.
  Interventions: Behavioral: Enhanced Usual Discharge Services-Residential

INTERVENTIONS:
Behavioral: Critical Time Intervention-Residential (CTI-R) — CTI-R is a 9-month, time-limited intervention that aims to produce an enduring impact by effectively linking individuals to both professional services (substance abuse and health and mental health providers) and social supports (e.g., family and friends) and by providing emotional and practical support. Participants in the CTI-R condition will also receive usual discharge services from the residential substance abuse treatment program.
  Arms: Critical Time Intervention-Residential
Behavioral: Enhanced Usual Discharge Services-Residential — The enhanced usual discharge condition encompasses the regular discharge services offered at the residential treatment program plus enhanced transition services.

SUMMARY:
This research uses a multi-phase approach to adapt and implement an established intervention, Critical Time Intervention, for a new population and setting among individuals with substance use who are at risk of relapse following residential substance abuse treatment. The goals of the study are to: (PHASE 1) identify challenges and strategies of community reentry among individuals in residential substance abuse treatment and their providers and social support networks (e.g., family, friends, community members); (PHASE 2) adapt CTI for individuals in residential substance abuse treatment to prepare them for discharge and transition back into the community; and (PHASE 3) conduct a pilot study to examine the feasibility, acceptability, and preliminary outcomes of the adapted CTI compared to enhanced usual discharge planning services.

DETAILED DESCRIPTION:
This randomized pilot study will examine the feasibility, acceptability, and preliminary outcomes of the adapted CTI compared to enhanced usual discharge planning services. More specifically, 60 participants will be randomized to either CTI (n=30) or enhanced usual discharge planning services (n=30) at the time of discharge. Participants will complete a baseline interview (prior to randomization) and 3-, 6-, 9- and 12-month follow-up assessments post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be enrolled in residential substance abuse treatment and who are at least 18 years of age, speak English, and expect to be discharged within 3 months.

Exclusion Criteria:

* Individuals that do not meet the aforementioned inclusion criteria will be excluded from the study.More specifically, the following categories will be excluded:

  1. Anyone under the age of 18
  2. Non-English speaking individuals due to limited resources
  3. Individuals who are considered vulnerable/protected populations, including children, pregnant women, and prisoners.
  4. Individuals judged by clinical treatment staff to be in immediate crisis, i.e., suicide watch or inadequate decisional capacity to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Enrollment | Baseline
  Proportion of participants enrolled in the study as measured by the research records
Change in retention | 3, 6, 9, and 12 months
  Proportion of participants completed the study as measured by the research records
Short-term Relapse | 3 months
  Proportion of participants who relapsed (i.e., substance use) as measured by Addiction Severity Index
Use of aftercare services | 3 months
  Proportion of participants who were linked to aftercare services (i.e. substance use treatment) at the time of discharge as measured by the Treatment Service Review (TSR)
Housing | 3 months
  Proportion of participants housed at the time of discharge

SECONDARY OUTCOMES:
Short-term Social Support | 3 months
  Level of social support as measured by the 8-item modified Medical Outcomes Study Social Support Survey
Short-term Self-Efficacy | 3 months
  Level of self-efficacy as measured by "I feel like I'm in control of my alcohol or drug use."
Short-term Mental Health | 3 months
  Level of mental health severity as measured by the Brief Symptom Inventory
Change in Relapse | 3, 6, and 9 months
  Proportion of participants who relapsed (i.e., substance use) as measured by Addiction Severity Index
Long-term Relapse | 12 months
  Proportion of participants who relapsed (i.e., substance use) as measured by Addiction Severity Index
Change in Social Support | 3, 6, and 9 months
  Level of social support as measured by the 8-item modified Medical Outcomes Study Social Support Survey
Long-term Social Support | 12 months
  Level of social support as measured by the 8-item modified Medical Outcomes Study Social Support Survey
Change in Self-Efficacy | 3, 6, and 9 months
  Level of self-efficacy as measured by "I feel like I'm in control of my alcohol or drug use."
Long-term Self-Efficacy | 12 months
  Level of self-efficacy as measured by "I feel like I'm in control of my alcohol or drug use."
Change in Mental Health | 3, 6, and 9 months
  Level of mental health severity as measured by the Brief Symptom Inventory
Long-term Mental Health | 12 months
  Level of mental health severity as measured by the Brief Symptom Inventory

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer I Manuel, PhD, Principal Investigator — New York University
Locations (1):
- New York University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No